CLINICAL TRIAL: NCT00328185
Title: Allograft Fibrosis: Its Regulation and Significance Following Pediatric Cardiac Transplantation
Brief Title: Allograft Fibrosis Following Pediatric Cardiac Transplantation
Status: Terminated | Type: Observational
Why Stopped: unable to gather sufficient data
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 05-217
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2006-01

CONDITIONS: Children Who Underwent Heart Transplantation Prior to Age 18; Received Care at Children's Healthcare of Atlanta
Keywords: pediatric; heart disease; orthotopic heart transplantation; allograft fibrosis
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Transplantation is the preferred method of treating many forms of end-stage organ failure. While short-term results have improved, long-term outcomes remain inadequate. Myocardial fibrosis could potentially have an adverse effect on long-term cardiac function. We wish to study the degree of fibrosis to see if we can predict survival following pediatric heart transplantation.

DETAILED DESCRIPTION:
There has been recent evidence that demonstrates a significant racial disparity in outcomes following pediatric heart transplantation.Differences in fibrosis or its regulation may offer an explanation to these differences.Just as the pathologic alterations of cardiac connective tissue in the ischemic heart and in cardiomyopathies support the view that the matrix plays a fundamental role in ventricular function,it is likely that other forms of cardiac dysfunction,such as that following heart transplantation,may also be related to changes in the extracellular matrix.Fibrosis has been identified in allografts following transplant,although the degree and significance relative to cardiac function remains unclear.Many of the regulatory substances have also been identified in the microenvironment of the allograft following transplant,but their role in collagen deposition and protease:anti-protease balance is unclear as well.It has been speculated that individual,racial,and regional disparities in outcome following pediatric heart transplantation may be the result of an underlying difference in fibrosis.This in turn influences the tolerance of the recipient to the graft,and ultimately,the time for graft failure to ensue.Of the 4227 pediatric heart transplants performed in the US 1987-2004,717 were African-American.The 1-year graft survival did not differ among groups;5-year graft survival was significantly lower among African-Americans compared to other racial groups.The median graft survival for African-American recipients was 5.3 years compared to 11.0 years for other recipients.African-American recipients had an increased likelihood of more HLA mismatches,lower median household income.After adjusting for disparities in a multivariate analysis, African-American race remained significantly associated with graft failure.While the cellular component of the myocardium has been extensively studied, the extracellular matrix is less well examined or understood.Processes of synthesis,degradation,and turnover are important for the understanding of the physiology of development and remodeling of tissues and the pathology of hypertrophy and fibrosis.Collagen Fibroblasts are responsible for the biosynthesis,assembly,and maintenance of the extracellular matrix. Collagen is one of the components of the extracellular matrix.While collagen proteins serve primarily as an inert structural support of connective tissue,they also control multiple cellular parameters such as adhesion,migration,cell shape,cytoskeletal architecture,and gene expression.Fibronectin is a protein of the extracellular matrix.Fibronectin primarily serves as an adhesive protein,facilitating cell adhesion to fibrin,collagens,heparin,and proteoglycans.Fibronectin is important in contact inhibition,cell movement,cell-substrate adhesion,inflammation,and wound healing.Another function of fibronectin may be in the homing of lymphocytic cells.Allograft rejection has been associated with infiltration of inflammatory cells and local deposition of fibronectin.Performing immunohistochemical analysis for collagen and fibronectin will determine the degree of fibrosis in serial endomyocardial biopsies over the duration of graft survival.This data will determine the correlation between allograft fibrosis and clinical parameters of cardiac function,and will uncover differences in the degree of fibrosis that may exist between racial groups.The interactions between cells,immune mediators,growth factors,and proteins that regulate fibrosis have been well documented in some clinical areas.Throughout the transplant literature,several points in the fibrosis cascade have been identified as potential important regulatory components. These include transforming growth factor-β,tumor necrosis factor-α,plasminogen activator inhibitor, matrix metalloproteinase-2,and matrix metalloproteinase-9.All have the possibility of affecting the production of collagen and fibronectin,and the degree of allograft fibrosis.Transforming growth factor-β has many properties.TGF-β has potential value as an immunosuppressant in tissue.It can serve as an anti-inflammatory agent based on its ability to inhibit the growth of both T and B cells.TGF-β has the ability to regulate growth depending on the surrounding cell type and whether or not other growth factors are present.TGF-β stimulates fibroblast chemotaxis and proliferation.As the most potent stimulator of collagen synthesis,it regulates deposition of extracellular matrix and cell attachment to it.It induces fibronectin,chondroitin/dermatin sulfate proteoglycans,collagen,and glycoaminoglycans.TGF-β promotes the formation and secretion of protease inhibitors,further contributing to collagen accumulation.TGF-β decreases collagenase,increases tissue inhibitors of metalloproteinases,and increases PAI-1 production.Studies have been done implicating TGF-β in the pathogenesis of small-airway fibrosis characteristic of obliterative bronchiolitis following lung transplant.TGF-β expression was higher in OB patients in comparison to patients without OB,and positive TGF-β staining preceded the histologic confirmation of OB by 6 months.TGF-β has been implicated as a contributing factor to the overproduction of collagen characteristic of dilated cardiomyopathy.Administration of neutralizing antibodies to TGF-β has been shown to limit collagen accumulation in wounds.Tumor necrosis factor-α is a cytotoxic monokine produced by macrophages. TNF-α is associated with the inflammatory response present following exposure to bacterial endotoxin.TNF-α is produced within the first three days of wound healing.It facilitates leukocyte recruitment,induces angiogenesis,and promotes fibroblast proliferation.In animal models,a prominent feature of acute allograft rejection is the dense deposition of fibronectin at the graft site.Administration of anti-TNF-α serum into the hosts abrogated acute rejection and prolonged allograft survival.It was accompanied by a decrease in intragraft TNF-α levels and down-regulated fibronectin mRNA expression.Certain serine proteases are thought to be key regulators of connective tissue turnover.Plasminogen activators generate plasmin,a serine protease,which has activity against a number of connective tissue macromolecules,including fibronectin,proteoglycan core proteins,other glycoproteins,collagen,as well as fibrin.Plasmin has been shown to initiate the autoactivation of other proteinases.The activity of plasminogen activators is closely regulated by specific inhibitors.The plasminogen activator inhibitors are potentially one of the most important regulators of connective tissue degradation because of their control of the rate of plasmin generation in local environments.PAI-1 is deposited pericellularly where its function is to regulate pericellular proteolysis.The connective tissue matrix metalloproteinase family consists of enzymes derived from mesenchymal cells and hematopoietic cells.They are metal-binding proteinases secreted in proenzyme forms requiring extracellular activation.The MMPs can be divided into subgroups,one of which is the interstitial collagenases.This group is responsible for regulating the extracellular collagen.Their activity is further regulated by a secreted inhibitor,tissue inhibitor of metalloproteinases,which forms a high-affinity irreversible complex with the active form of the MMP.Whether or not matrix production and degradation occur depends on the relative amounts of the metalloproteinases and inhibitors and also on the complex interplay with serum inhibitors.In disease states where the control mechanisms become uncoordinated,the uaction and nature of MMP activities may be one of the factors leading to an imbalance of the extracellular matrix.Studies have shown an increased expression of several MMPs during cardiac,renal,and pulmonary allograft rejection.In animals,allografts in the presence of MMP-9 showed lower cellular infiltration and fibrosis than allografts harvested from MMP-9 deficient recipients.The reverse was true with MMP-2,suggesting that MMP-2 and MMP-9 may play different roles in the process of allograft fibrosis and rejection.By performing immunohistochemical analysis,we will determine the various amounts of these potential regulatory substances in serial endomyocardial biopsies over the duration of graft survival.This data will allow us to compare the changes in regulatory factors with the degree of fibrosis over time.It will enable us to uncover differences in regulation that may exist between racial groups.During the isovolumetric contraction phase of systole,ventricular wall pressure develops rapidly.During the ejection phase,pressure is transmitted to the ventricular cavity.Associated with ejection,geometric changes occur in the ventricle.Transmission of force to the ventricle must involve the myocardial matrix.Of the structural proteins in the heart,collagen has the physical properties necessary for force transmission to the ventricle.One can conclude that a complex system composed primarily of collagen is necessary for at least systolic stress distribution and tethering of myocytes one to another during the spatial translocations that accompany systole.For proper ventricular function,contiguous myocytes must be stretched to near the same amount.This implies a mechanism for distribution of stress throughout the entire ventricular wall.It appears that not only the total amount or collagen present,but also the distribution may be important.Increases and decreases in collagen have been noted in various disease states and affect cardiac function.The pathologic alterations of the intrinsic cardiac connective tissue in the ischemic heart and in cardiomyopathies support the view that the extracellular matrix plays a fundamental role in ventricular function.Ischemic damage of the myocardium is a blood flow-mediated,time-dependent process.Even in the absence of tissue necrosis,there is reversible loss of contractile function.Although myocytes are not morphologically damaged when stunned,they may lose their interconnections through damage to collagen and the extracellular matrix.The individual cells then move relative to each other without generating coordinated,forceful contractions.In animals,studies have shown systolic bulging,mural thinning,and regions of absent connective tissue.With congestive cardiomyopathy,there is ventricular dilation,global wall thinning and diffuse contractile dysfunction.Although a significant component of ventricular dysfunction may relate to loss of contractile mass,there are regions of connective tissue absence within the normal myocardium in animal models.The untethering of myocytes again leads to defective,uncoordinated contractile activity.Similarly,the loss or damage of intrinsic connective tissue may account for the characteristic global wall thinning.This may lead to a spiral of progressive damage;as the ventricular cavity enlarges,end-diastolic pressure increases,thereby causing further injury to the connective tissue.In contrast to congestive cardiomyopathy,some forms of heart disease are associated with decreased compliance and diminished diastolic filling.Increased collagen has been demonstrated in hypertrophied hearts.Rather than a thin-walled dilated heart,animal models demonstrate mural hypertrophy with a small ventricular cavity.In patients with hypertrophic,obstructive cardiomyopathy,biopsies of the septum revealed severe myocellular hypertrophy,myocyte disorganization,and pronounced interstitial collagen deposition.There is an increase in all components and disorganization in the arrangement.After quantifying the degree of fibrosis and the various amounts of regulatory substances,we will correlate this data to clinical parameters.We will compare changes in fibrosis over time with measurements of cardiac function,and with graft survival.

ELIGIBILITY:
Inclusion Criteria:

* Children who underwent heart transplantation prior to age 18
* Followed up at Children's Healthcare of Atlanta

Exclusion Criteria:

* Children without a transplanted heart
* Follow-up not at children's Healthcare of Atlanta

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who underwent heart transplantation prior to age 18
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2006-01; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian E Kogon, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States